CLINICAL TRIAL: NCT04548011
Title: Acupuncture of Different Treatment Frequency on Improving Quality of Life in Patients With Functional Dyspepsia: a Three-armed Randomized Controlled Trial
Brief Title: Acupuncture of Different Treatment Frequency on Improving Quality of Life in Patients With Functional Dyspepsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Biyun Sun, Department of Acupuncture doctor in Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAMHospital20200906
Record Dates: First submitted 2020-09-06; First posted 2020-09-14 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Three times a week group (Experimental): Twenty participants in three times a week group will receive acupuncture treatment 3 times per week (every other day) for 4 weeks, 12 sessions totally. The acupuncture operation as above. Participants will not be not allowed to take any other medication or accept any treatment for FD. should not be accepted during the study. In case of unbearable symptoms, the assistant researchers will detailly document.
  Interventions: Other: Acupuncture
- Once a week group (Experimental): Twenty participants in once a week group will receive acupuncture treatment 1 time per week for 4 weeks (Weekly fixed day), 4 sessions totally. Other inventions will be same as the Three times a week group.
  Interventions: Other: Acupuncture
- Waiting for treatment group (No Intervention): After the health education（such as dietary adjustment for FD patients）, the participants will be followed up for 4 weeks. At the end of the follow-up, the patients could be given free acupuncture treatment (the invention will be similar with that of the Three times a week group) for 4 weeks at will.

INTERVENTIONS:
Other: Acupuncture — The acupuncture treatment strategies in this study are based on traditional Chinese medicine theory and opinions from the acupuncture experts. The acupoints are bilateral Zhongwan（CV12）, Tianshu（ST25）, Neiguan（PC6）, Liangqiu（ST34）, Yanglinquan（GB34）, Zusanli（ST36）and Taichong（LR3）.All the acupoints will be localized according to the Nomenclature and Location of Acupuncture Points of the People's Republic of China. During the acupuncture treatment, the participants will be in supine position. After 75% alcohol pads sterilizing the skin around the acupoints routinely, the acupuncturists will use sterile disposable steel needles (0.3 mm×40 mm; Huatuo Brand, Suzhou Medical Appliance, China) to insert into the acupoints above. The acupoints will be inserted vertically at 13-40 mm with the manipulation of steady small lifting, thrusting, and twirling 3 times to induce a sensation of de qi (sourness, numbness, and heaviness).
  Arms: Once a week group; Three times a week group

SUMMARY:
The objective of this trial is to assess acupuncture of different treatment frequency on improving quality of life in patients with functional dyspepsia.

DETAILED DESCRIPTION:
The effect of treatment frequency of acupuncture on the functional dyspepsia is unclear. In this study, 60 participants with FD will be recruited and randomly allocated (using a 1:1:1 allocation ratio) into three times a week group, once a week group and waiting for treatment group. Participants will receive acupuncture treatment at bilateral Zhongwan（CV12）, Tianshu（ST25）, Neiguan（PC6）, Liangqiu（ST34）, Yanglinquan（GB34）, Zusanli（ST36）and Taichong（LR3) of different treatment frequency for 4 weeks. This trial is designed to analyze the acupuncture of different treatment frequency on improving quality of life in patients with FD and to provide evidence for the establishment of acupuncture treatment quantization standard of FD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of FD as defined by the Roman IV Functional Dyspepsia Diagnostic criteria

   One or more of the following:
   1. Bothersome postprandial fullness
   2. Bothersome early satiation
   3. Bothersome epigastric pain
   4. Bothersome epigastric burning AND No evidence of structural disease (including at upper endoscopy) that is likely to explain the symptoms Epigastric Pain Syndrome (EPS) criteria: fulfilled for the last 3 months with symptom onset at least 6 months before diagnosis.

   Postprandial Distress Syndrome Diagnostic (PDS) criteria: must include one or both of the following at least 3 days per week:
2. Age 18-75 years.
3. Signed informed consent and volunteered to participate in the trial.

Exclusion Criteria:

Candidate participants with any of the following items will be excluded from this trial.

1. Gastrointestinal motility drugs taken within the past 15 days; Acupuncture treatments within the past 30 days; participating in other ongoing clinical trials
2. Severe heart, lung, liver, brain or kidney damage.
3. Would-be mothers, pregnant or lactation;
4. Progressive malignant tumor or other severe consumptive diseases, easy to be complicated with bleeding and infection;
5. Cognitive impairment such as unable to express subjective symptoms of discomfort or give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The score change in Nepean Dyspepsia Life Quality Index compared with baseline at week 4 | week 4
  The primary outcome is the score change in Nepean Dyspepsia Life Quality Index （NDLQI）compared with baseline at week 4. The NDLQI is a scale of 25 items about the quality of the patients' life with a ranging score of 1-4 of each item. The higher scores indicates a worse outcome.

SECONDARY OUTCOMES:
The score change in NDLQI compared with baseline | week 2, week 8 and week 12
  The score change in NDLQI compared with baseline at weeks 2, 8 and 12. The NDLQI is a scale of 25 items about the quality of the patients' life with a ranging score of 1-4 of each item. The higher scores indicates a worse outcome.
The score of each dimension change in NDLQI compared with baseline | week 4, week 8 and week 12
  The score of each dimension change in NDLQI compared with baseline at weeks 4, 8 and 12. The NDLQI is a scale of 25 items about the quality of the patients' life with a ranging score of 1-4 of each item. The higher scores indicates a worse outcome.
The total score change in Symptom Index of Dyspepsia （SID） | week 4, week 8 and week 12
  The total score change in Symptom Index of Dyspepsia （SID） compared with baseline at weeks 4, 8 and 12. SID is a four-rate scale with a ranging score of 0-4 of each dyspepsia symptoms (postprandial distension; early satiety; epigastric pain; and epigastric burning). The higher scores indicates a worse outcome.
The standard score change in Self-Rating Anxiety Scale（SAS） | week 4, week 8 and week 12
  The standard score change in Self-Rating Anxiety Scale（SAS） compared with baseline at weeks 4, 8 and 12. SAS is a scale of 20 items about the anxiety level of patients with a ranging score of 1-4 of each question. The higher scores indicates a worse outcome.
6. The standard score change in Self-Rating Depression Scale （SDS） | week 4, week 8 and week 12
  The standard score change in Self-Rating Depression Scale （SDS） compared with baseline at weeks 4, 8 and 12. SAS is a scale of 20 items about the depression level of patients with a ranging score of 1-4 of each question. The higher scores indicates a worse outcome.